CLINICAL TRIAL: NCT04775017
Title: Delirium in Covid-19: Germany-wide Covid-19 Intensive Register
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: COVID-19-Delirium
Record Dates: First submitted 2021-01-21; First posted 2021-03-01 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Intensive Care Unit Delirium; Covid19; Post Intensive Care Unit Syndrome
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The global pandemic caused by the SARS-CoV-2 virus is confronting the German health system with a novel pathogen. This means that a timely evaluation of all available results is required. In the field of intensive care in particular, there are significant gaps in knowledge, particularly with regard to delirium. In this respect, this study also serves directly to investigate the pathways of delirium outcome in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

All patients with SARS-CoV-2 positive Covid-19 disease

* Age≥18 years
* Proven by positive PCR tests from nasal/ throat swabs as well as samples from the deep respiratory tract.
* Period 01.01.2020 to 21.02.2022

Exclusion Criteria:

* NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have COVID-19 and have been treated in an intensive care unit of Charité Universitätsmedizin and whose therapy has already been completed on 21.02.2022.
Sampling Method: Probability Sample
Enrollment: 2398 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | 01.01.2020 - 21.02.2022
  Delirium is measured by validated screening scores.

SECONDARY OUTCOMES:
Risk factors for severe COVID-19 | 01.01.2020 - 21.02.2022
  Risk factors are defined according to actual literature e.g. obesity, diabetes or hypertension.
Patient characteristics | 01.01.2020 - 21.02.2022
  Patient characteristics at hospital admission e.g. score level
Blood gas analysis | 01.01.2020-31.07.2020
  Monitoring of blood gas analysis
Enteral nutrition | 01.01.2020-31.07.2020
  Monitoring of enteral nutrition
Parenteral nutrition | 01.01.2020 - 21.02.2022
  Monitoring of parenteral nutrition
Serum albumin | 01.01.2020 - 21.02.2022
  Monitoring of serum albumin level
Total protein | 01.01.2020 - 21.02.2022
  Monitoring of total protein level
Phosphate | 01.01.2020 - 21.02.2022
  Monitoring of phosphate levels
Triglyceride | 01.01.2020 - 21.02.2022
  Monitoring of triglyceride levels
Caloric intake | 01.01.2020 - 21.02.2022
  Caloric intake is measured by total daily energy supply.
Respiratory setting | 01.01.2020 - 21.02.2022
  Respiratory factors are measured respiratory setting
Inflammatory laboratory parameter 1 | 01.01.2020 - 21.02.2022
  Monitoring of interleukine level
Inflammatory laboratory parameter 2 | 01.01.2020 - 21.02.2022
  Monitoring of cytokine level
Inflammatory laboratory parameter 3 | 01.01.2020 - 21.02.2022
  Monitoring of big immune status
Inflammatory laboratory parameter 4 | 01.01.2020 - 21.02.2022
  Monitoring of t-cell population
Toxic-drug factors | 01.01.2020 - 21.02.2022
  Toxic-drug factors are measured by concomitant medication.
Sociodemographic factors | 01.01.2020 - 21.02.2022
  Sociodemographic factors are measured by Audit, Fagerström, occupation, age, gender, cognitive status.
Breathing hours | 01.01.2020 - 21.02.2022
  Breathing hours are measured by non-invasive and invasive ventilation.
Length of intensive care unit stay | 01.01.2020 - 21.02.2022
  Length of intensive care unit stay is measured in days of stay in the intensive care unit.
Length of hospital stay | 01.01.2020 - 31.07.2022
  Length of hospital stay is measured in days of stay in hospital.
Adverse events | 01.01.2020 - 21.02.2022
  Adverse Events defined by thromboembolic events, nosocomial infections, septic shock, acute renal failure, heart attack, post-intensive care syndrome and death are recorded until hospital discharge.
Post Intensive Care Unit Syndrome (PICS) | 01.01.2020 - 21.02.2022
  Post Intensive Care Unit Syndrome (PICS) is measured by a validated battery (composite endpoint).
In-hospital mortality | 01.01.2020 - 21.02.2022
  Mortality is measured in the hospital
Mortality | 01.01.2020 - 31.08.2022
  Mortality is measured until 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charité - Universitäsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine Campus Virchow-Klinikum, Berlin, Germany